CLINICAL TRIAL: NCT06933394
Title: A Prospective, Single-arm, Multicentre Phase II Clinical Study of Arsenic Trioxide in Combination With Chemotherapy and MAPK Pathway Inhibitors for Stage 4/M Neuroblastoma
Brief Title: Arsenic Trioxide With MAPK Inhibitors and Chemotherapy for Stage 4/M Neuroblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-749-02
Record Dates: First submitted 2025-02-07; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; arsenic trioxide; MAPK inhibitor
MeSH Terms: conditions — Neuroblastoma | interventions — Arsenic Trioxide; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experiment group (Experimental)
  Interventions: Drug: Arsenic trioxide; Drug: MAPK inhibitors; Drug: Chemotherapy

INTERVENTIONS:
Drug: Arsenic trioxide — Patients will receive 9 cycles of chemotherapy. ATO dosing: Arsenic trioxide（ATO） is administered 0.18mg/kg per day over eight hours IV daily for ten days. Patients will receive ATO alone on days 1-2 and combined with conventional induction chemotherapy on days 3-10.
Drug: MAPK inhibitors — The dosage of MAPK inhibitors is adjusted based on the specific drug. For example, Trametinib is used as follows: Trametinib will be administered daily from Cycle 5 until the end of induction chemotherapy. Patients start at Dose Level I; if no hematologic toxicity or severe drug-related complications occur after 1 cycle, the dose is escalated to the next level, otherwise, it is maintained. Dose Level I: 0.016 mg/kg/day (<6 years) or 0.012 mg/kg/day (>6 years), po. qd. Dose Level II: 0.024 mg/kg/day (<6 years) or 0.018 mg/kg/day (>6 years), po. qd. Dose Level III: 0.032 mg/kg/day (<6 years) or 0.025 mg/kg/day (>6 years), po. qd.
  The dosages of other MAPK inhibitors should be modified according to their respective recommended therapeutic guidelines.
Drug: Chemotherapy — The conventional chemotherapy regimens are as follows:
  Cycles 1, 2, 4, and 6 follow the CAV regimen (cyclophosphamide(1.2g/m2.d, d3-d4), pirarubicin(25mg/m2.d,d3-d5), vincristine(0.022mg/kg.d or 0.67mg/m2.d，d3-d5)).
  Cycles 3, 5, and 7 follow the PVP regimen (cisplatin(50mg/m2.d, d3-d6), etoposide(200mg/ m2.d, d3-d5)).
  Cycles 8 and 9 follow the CT regimen (cyclophosphamide(1.2g/m2.d, d3-d4), topotecan(2mg/m2.d, d3-d5)).

SUMMARY:
This prospective, single-arm, multi-center clinical trial aims to explore and evaluate the efficacy and safety of the combination therapy involving arsenic trioxide, MAPK inhibitors, and chemotherapy for stage 4/M neuroblastoma.

DETAILED DESCRIPTION:
Neuroblastoma (NB) is the most common extracranial solid tumor in children. Since 2018, we have led a prospective, nationwide multicenter collaborative clinical study on arsenic trioxide(ATO) combined with chemotherapy for 4/M stage NB (NCT03503864).The results indicate that the objective response rate (ORR) and complete remission rate (CRR) at the end of induction (EOI) for the ATO-combined chemotherapy regimen are significantly higher than those of the commonly used NB regimens in China, as well as the internationally recognized rCOJEC and MSKCC-N5 regimens. Additionally, the ATO regimen demonstrates a lower incidence of toxic side effects, providing favorable conditions for subsequent consolidation therapy and contributing to the long-term survival of High-risk neuroblastoma(HR-NB) patients. However, in clinical practice, we found that some children responded poorly to ATO combined induction chemotherapy, with lesions persisting or progressing and recurring, gradually developing into refractory cases during induction chemotherapy. Studies show that primary/acquired resistance in NB is related to the high-frequency clonal diversity that gradually emerges with chemotherapy.

With the advancement of precision medicine technology and in-depth research on signaling pathways, we found the RAS-MAPK signaling pathway plays an important role in the regulation of cell proliferation and differentiation, and this pathway is abnormally activated in various tumors. Literature reports that 78% of refractory/recurrent NB have activating mutations in the RAS-MAPK pathway, suggesting a close association between this pathway and refractory/recurrent NB. In addition, in some tumor cell lines, ATO can cause upregulation of the MAPK pathway, which may be the reason for the poor efficacy of ATO in some HR-NB children and suggests the necessity of combining MAPK inhibitors in ATO-containing induction chemotherapy regimens. Studies have shown that in APL cell line NB4 and APL primary cells, MAPK (MEK) inhibitors (PD98059 and PD184352) enhance apoptosis in ATO-treated cells by inhibiting downstream ERK1/2 and Bad phosphorylation, indicating that combining ATO with MAPK inhibitors can further improve efficacy.

Clinical studies show that single-agent MAPK inhibitors often have poor efficacy in the treatment of advanced or refractory tumors. Studies have found that in ALK-dependent RAS-MAPK mutant NB cell lines, MAPK inhibitors can activate the pro-cancer PI3K-AKT pathway through the mTORC2 complex-related subunit SIN1, and thus the MAPK inhibitor trametinib cannot inhibit the growth of ALK-dependent NB in mouse models. Previous studies have found that ATO can downregulate the PI3K-AKT pathway in various tumors, and we have found through non-label quantitative proteomics technology that ATO treatment of NB cell line SK-N-BE(2) can also cause downregulation of this pathway, and studies have shown that ATO can inhibit the activity of the mTORC2 complex in this pathway. In summary, we propose combining ATO with MAPK inhibitors, with the aim of using MAPK inhibitors to counteract the adverse effects of ATO activating the MAPK pathway, while ATO inhibits the activation of the PI3K-AKT pathway caused by MAPK inhibitors, thereby jointly inhibiting tumor growth.

As chemotherapy progresses, tumor cells gradually accumulate DNA damage under chemotherapy pressure, leading to a higher probability of gene mutations and clonal evolution associated with poor prognosis, increasing the likelihood of drug resistance; studies show that primary/acquired resistance in NB is also related to the high-frequency clonal diversity that gradually emerges with chemotherapy; under the selective pressure of chemotherapeutic drugs, cells with drug-resistant characteristics gradually expand and enrich, and gradually dominate; the later the remission time during induction chemotherapy in NB patients, the worse the prognosis; studies show that patients with initial bone marrow minimal residual disease(MRD) positivity who remain positive after 4 courses of chemotherapy have a significantly higher recurrence rate than those who become negative (74.1% vs. 33.3%), and the event-free survival has statistical significance; and radical surgery performed after the 3rd or 4th course of induction chemotherapy according to consensus and mainstream cooperative group regimens may also be one of the potential risk factors promoting the dissemination and metastasis of NB tumor cells; therefore, we chose to add trametinib to the medication sequence starting from the 5th course of induction chemotherapy, for a total of 5 courses of combined medication (the 5th to 9th courses of induction chemotherapy). The effectiveness and safety of the above combined medication strategy need to be further verified through multicenter collaborative clinical studies, and we expect that this combined medication regimen can improve the treatment status and prognosis of HR-NB, a refractory tumor.

Based on the above theoretical basis, the combination of MAPK pathway inhibitors with ATO has a synergistic effect, and we expect that the new regimen of adding the MAPK pathway inhibitor trametinib to the original ATO combined chemotherapy regimen can improve CRR. Therefore, this study aims to use the CRR at EOI of ATO combined chemotherapy and MAPK signaling pathway inhibitor(for example. trametinib) in the treatment of 4/M stage NB as the main research objective. The overall CRR at EOI for 4/M stage NB, both domestically and internationally, will serve as an external control to assess the clinical efficacy and safety of ATO-combined chemotherapy plus the MAPK signaling pathway inhibitor during the induction chemotherapy phase of 4/M stage NB.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of neuroblastoma.
2. Preoperative staging as INRG M stage or postoperative staging as INSS stage 4 (regardless of risk classification).
3. Age ≥18 months and ≤18 years.
4. Informed consent obtained from the legal guardian, and signed informed consent form.

Exclusion Criteria:

1. Patients with a history of other tumors who have received chemotherapy and abdominal radiation therapy.
2. Severe progressive or persistent heart failure: NYHA heart function class III or IV, or left ventricular ejection fraction (LVEF) < 50%.
3. Severe progressive or persistent renal failure: glomerular filtration rate (GFR) < 30 ml/(min·1.73 m²) or serum creatinine > 5 mg/dL (442 μmol/L).
4. Severe liver dysfunction: aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≥ 5× upper limit of normal (ULN), or serum total bilirubin ≥ 3× ULN.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2031-05-01 (Estimated); Study Completion 2031-05-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CRR) | Four weeks after ATO-combined chemotherapy
  Complete remission rate

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Four weeks after ATO-combined chemotherapy
  Objective Response Rate
Disease Free Survival | 3 years
  The proportion of patients who have not experienced recurrence of disease or death from any cause, whichever occurs first, within a maximum of 3 years from the date of enrollment.
Overall survival | 3 years
  The proportion of patients who are alive from the date of randomization to 3 years, regardless of the cause of death.
Incidence of Adverse Events | From the start of the combined regimen until the first documented adverse event, up to 3 years.
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided